CLINICAL TRIAL: NCT02727920
Title: A Test of the Effects of Energy Drinks
Brief Title: Effects of Energy Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 00006831
Record Dates: First submitted 2016-03-26; First posted 2016-04-05 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Energy Drinks
MeSH Terms: interventions — Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): drink containing pyridoxine, folate; B12); taurine, choline, glucuronic acid; tyrosine, phenylalanine*, malic acid, and caffeine administered one time.
  Interventions: Dietary Supplement: Energy drink
- Placebo drink (Placebo Comparator): Placebo drink administered one time.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Energy drink
  Arms: Experimental
Other: Placebo — placebo drink
  Arms: Placebo drink

SUMMARY:
This study is designed to test the efficacy of energy drinks. This is a double-blinded, crossover, randomized clinical trial, measuring the effect of the test drinks compared with placebo drink in 200 participants aged 18-70 years.

DETAILED DESCRIPTION:
This study is designed to test the efficacy of an energy drink compared to placebo via a double-blind, crossover, randomized clinical trial. Energy levels will be assessed before and after consumption of the test beverages on 2 days separated by a week in 200 participants aged 18-70 years. The study is crossover because the participants will be (randomly) receiving one drink on Test Day 1 and the other drink on Test Day 2.

After signing written informed consent, participants will be fed a light lunch, and their pulse, weight and height measured. A baseline battery of computer-based tests to assess energy levels will be conducted. These computer-based measures will take ~40 minutes to complete and will include: a) a long-term memory test b) a Profile of Mood States (POMS2) brief form; c) Rapid Visual Information Processing (RVIP) test, d) The N-Back Task; d) Reaction time online test; f) the Flanker Task. Participants will then be asked to fill out a baseline survey (30 min), with questions about current health-related behaviors, specifically questions about physical activity and diet.

Upon completing the baseline battery (survey administered at test session 1 only), participants will be randomly administered the energy drink or the placebo to consume while observed. Subsequently, the battery of computer-based tests to assess energy levels will be re-administered 30 minutes, 2.5 hours and 5 hours after consumption of the test drink.

The study intervention will be double-blinded: participants will be blinded to whether they are receiving the active or the placebo drink, and study team members will also not be aware of the assignment.

When the study ends, full compensation will be given if the intervention is fully completed; if the intervention is not fully completed, partial compensation will be given.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in reading English
* High school graduate as lowest education level

Exclusion Criteria:

* Non-smoker
* No diagnosed/treated cognitive/psychiatric conditions by self-report
* No diagnosed/treated diabetes, hypoglycemia or thyroid condition by self-report
* No current use of prescription stimulant medications by self-report
* No allergies or sensitivities to foods, ingredients or chemicals by self-report, that are contained in the test drink or placebo
* No diagnosed phenylketonuria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2016-04-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
attention-memory score | 5 hours
  Comparing intervention to placebo results on attention-memory score

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burrows T, Pursey K, Neve M, Stanwell P. What are the health implications associated with the consumption of energy drinks? A systematic review. Nutr Rev. 2013 Mar;71(3):135-48. doi: 10.1111/nure.12005. Epub 2013 Jan 29. PMID 23452281
- [Background] Goldfarb M, Tellier C, Thanassoulis G. Review of published cases of adverse cardiovascular events after ingestion of energy drinks. Am J Cardiol. 2014 Jan 1;113(1):168-72. doi: 10.1016/j.amjcard.2013.08.058. Epub 2013 Oct 4. PMID 24176062
- [Background] Ali F, Rehman H, Babayan Z, Stapleton D, Joshi DD. Energy drinks and their adverse health effects: A systematic review of the current evidence. Postgrad Med. 2015 Apr;127(3):308-22. doi: 10.1080/00325481.2015.1001712. Epub 2015 Jan 6. PMID 25560302
- [Background] Rath M. Energy drinks: what is all the hype? The dangers of energy drink consumption. J Am Acad Nurse Pract. 2012 Feb;24(2):70-6. doi: 10.1111/j.1745-7599.2011.00689.x. Epub 2012 Jan 31. PMID 22324861
- [Background] Kurtz AM, Leong J, Anand M, Dargush AE, Shah SA. Effects of caffeinated versus decaffeinated energy shots on blood pressure and heart rate in healthy young volunteers. Pharmacotherapy. 2013 Aug;33(8):779-86. doi: 10.1002/phar.1296. Epub 2013 May 30. PMID 23722481
- [Background] Phan JK, Shah SA. Effect of caffeinated versus noncaffeinated energy drinks on central blood pressures. Pharmacotherapy. 2014 Jun;34(6):555-60. doi: 10.1002/phar.1419. Epub 2014 Mar 19. PMID 24644139
- [Background] Shah SA, Nguyen NN, Bhattacharyya M. Energy Implications of Consuming Caffeinated Versus Decaffeinated Energy Drinks. J Pharm Pract. 2015 Oct;28(5):482-3. doi: 10.1177/0897190015585738. No abstract available. PMID 26378195
- [Derived] Garcia-Alvarez A, Cunningham CA, Mui B, Penn L, Spaulding EM, Oakes JM, Divers J, Dickinson SL, Xu X, Cheskin LJ. A randomized, placebo-controlled crossover trial of a decaffeinated energy drink shows no significant acute effect on mental energy. Am J Clin Nutr. 2020 Mar 1;111(3):719-727. doi: 10.1093/ajcn/nqz343. PMID 31990972